CLINICAL TRIAL: NCT01350453
Title: Development and Pilot Evaluation of a Web-supported Programme of Constraint Induced Therapy Following Stroke (LifeCIT)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Southampton (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); University Hospital Southampton NHS Foundation Trust (Other); Royal Bournemouth and Christchurch Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Jane Burridge, PhD, Professor, University of Southampton
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PB-PG-0909-20145
Record Dates: First submitted 2011-05-06; First posted 2011-05-09 (Estimated); Results first posted 2019-05-06 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-02

CONDITIONS: Stroke
Keywords: CIT; Stroke
MeSH Terms: conditions — Stroke | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LifeCIT (Experimental): Participants will be asked to aim to wear the C-MIT for 9 hours a day for 5 days/week, including 4-6 hours of structured activities per day: two 30-60 minute sessions of web-based activities and 3-4 hours practicing everyday activities.
  Interventions: Behavioral: LifeCIT
- Standard Care (Active Comparator): Participants received their usual care which included home exercises
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: LifeCIT — Participants will be asked to aim to wear the C-MIT for 9 hours a day for 5 days/week, including 4-6 hours of structured activities per day: two 30-60 minute sessions of web-based activities and 3-4 hours practicing everyday activities.
  Arms: LifeCIT
Behavioral: Standard Care — Participants will receive their usual care from their NHS provider.
  Arms: Standard Care

SUMMARY:
When a person has had a stroke they often lose their confidence, motivation and the ability to move one arm and hand. Recent research has shown that intensive exercise assists recovery of movement, but people are often discouraged by slow progress and stop using their weak limb.

A new idea, called Constraint Induced Therapy (CIT), has been shown to overcome this habitual 'non-use'. CIT involves wearing a mitt on the unaffected hand for several hours a day to prevent it from being used. Use of the weak arm and hand is encouraged by intensive exercises. CIT is not available in the NHS because of lack of therapist time for supervision and patients lack the confidence and motivation to carry out CIT alone at home.

This study will have two stages.

Stage 1.

The aim of this part of the study is to develop a web-based therapy programme ('LifeCIT') to support patients carrying out CIT at home (with their carer where possible) with online therapist support. The investigators will develop the therapy programme working closely with at least 12 patients, 6 carers and 6 therapists to identify and resolve any problems.

Stage 2

The investigators will then carry out a pilot trial in 6 treatment centers with 20 patients who have just been discharged from hospital and who have loss of arm and hand function. To test LifeCIT the investigators will randomly allocate patients to receive either the LifeCIT intervention or usual care. A researcher, who doesn't know which group patients have been allocated to, will measure their arm and hand function, record the problems this causes and how it affects their quality of life. Tests will be repeated after treatment (3 weeks) and 6 months later. The investigators will also examine the cost-effectiveness of treatment and ask both therapists and patients for their views.

DETAILED DESCRIPTION:
Development and pilot evaluation of a web-supported programme of Constraint Induced Therapy following stroke (LifeCIT) PB-PG-0909-20145

Jane H. Burridge PhD1, Claire Meagher MSc1, Ann-Marie Hughes PhD1, Sean-Ewings PhD2, Ana-Carolina Gonçalves BSc1, Claudia H. S. Alt PhD1, Sebastien Pollet BSc1, Lucy Yardley PhD3

1. Rehabilitation and Health Technologies Research Group, Faculty of Health Sciences, University of Southampton, United Kingdom.
2. Faculty of Statistical Sciences, University of Southampton, United Kingdom.
3. Faculty of Health Psychology, University of Southampton, United Kingdom.

Lay Summary

Background:

Following stroke people often lose their motivation and ability to move their hemiplegic arm. Intensive exercise assists recovery, but people often get into the habit of not using their arm.

Constraint-Induced Therapy (CIT) overcomes this habitual 'non-use'. CIT involves wearing a mitt on the unaffected hand to prevent it from being used. Use of the weak arm is encouraged by intensive exercises. CIT is not generally available in the NHS because of lack of therapist time to supervise the intensive exercises. We found that patients lack the confidence and motivation to carry out CIT alone at home.

We developed a web-based therapy programme ('LifeCIT') to support patients carrying out CIT at home with online therapy support. We developed LifeCIT working closely with patients, their carers and therapists. Their feedback and ideas ensured LifeCIT satisfied their needs. The first working version of LifeCIT was tested with 12 patients who had recently had a stroke and their feedback was used to make further improvements. A pilot trial with 19 patients tested whether LifeCIT affected recovery. We randomly allocated each patient to receive either 'LifeCIT' or 'usual care'. We tested patients before the study and repeated measurements after treatment (3 weeks) and 6 months later. We asked the patients who had used LifeCIT for their views on it - what was good and bad, and whether it had affected their ability to use their arm and hand.

Summary of research

Background:

Conventional therapy to improve upper limb function following stroke is not effective. <50% of people who survive a stroke but have moderate to severe hemiparesis regain upper limb function. Learnt non-use has been identified as an important factor in poor recovery. Constraint-Induced Therapy (CIT) [1; 2], proposes that constraint of the unaffected arm and hand, coupled with intensive training of the hemiplegic limb, leads to behavioral changes towards greater use of the hemiplegic limb, neuroplastic cortical changes and the return of function [3].

Despite evidence from a large RCT (n=222), which showed improvement in function maintained at 12 months post-treatment [4], CIT has not translated into clinical practice, due partly to the cost of intensive (minimum 4 hours/day for 10 days) one-to-one treatment. An alternative approach in which CIT was used at home without intensive therapy showed in an A-B-A trial, but patients reported lack of motivation to wear the C-MIT (Constraint Mitt) and comply with the exercise programme [5].

LifeGuide is a set of software resources to create and modify programmes of personalized online support for therapy, without the need for costly dedicated programming. It was used in this study to address the motivational barriers to home-based CIT.

Aims and Objectives:

1. Working with patients, carers and therapists, create an accessible and engaging web-supported programme of CIT for home-based upper limb stroke rehabilitation - LifeCIT.
2. Conduct a Phase II single-blinded RCT of LifeCIT to:

   1. Generate preliminary data on the effect size of the intervention compared with usual care for the purposes of calculating the power of a future phase III trial.
   2. Assess patients' views and adherence to the intervention and identify issues affecting the acceptability and feasibility of implementing and trialing the LifeCIT intervention.

Methods:

Phase 1. Intervention development:

The LifeCIT web-based programme for CIT combined with personalized activities, automated progress-relevant advice intervention content and format was co-designed with patients, carers and healthcare professionals. We held a series of meetings in which participants were shown mock-up webpages. Pages, structure, content, and activities were revised through a systematic response to feedback and then further revisions were made through in-depth think-aloud sessions with four chronic stroke patients.

During the development, process tape-recorded interviews and observational ('think aloud') studies [6-8] were used. Data collection and analysis was concurrent with intervention development, allowing immediate modification and re-testing of intervention components as potential improvements were identified.

The prototype web-based programme was then trialed with 12 sub-acute patients and their carers/ healthcare professionals and further revisions were made. The final version of the web-support programme was designed to:

1. Provide personalized treatment protocols (including targets for C-MIT wearing, web-based repetitive and functional activities). The patient was encouraged to log-on each morning to plan a programme of C-MIT wearing and activities and to complete a set of repetitive exercises. They were asked to log-on again later in the day to report on adherence to the activities, any difficulties encountered, and to complete the second set of repetitive exercises.
2. Provide structured support on progress and activities and automated support, based on activities and performance, including reminders (e.g. email or text messages to the patient and/or carer); motivational messages and suggestions for overcoming barriers.

Phase II Clinical trial:

A 6-center 3-week pilot trial compared usual care with LifeCIT. Computer block-randomization stratified into three ability groups. Participants randomized to the LifeCIT group were asked to wear the C-MIT for between 6 and 9 waking hours and aim for up to 6 hours activities per day on 5 days/week. A programme of activities was designed with them.

Participants Two cohorts of participants were recruited: One, sub-acute patients following discharge from hospital and one of the participants who had experienced a stroke more than 16 weeks previously.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ischaemic or haemorrhagic stroke affecting either right or left upper limb
* Either: a) Able to transfer safely between toilet, chair and standing and able to walk safely at home wearing the C-MIT with or without the use of a walking aid or b) primarily a wheelchair user having help or supervision to transfer and walk
* Mini-mental score >23
* Minimum of 10 degrees of active wrist extension measured by a hand held goniometer
* Discharged home from hospital (not institutional care)
* Access to internet at home

Exclusion Criteria:

* Major medical problems that could interfere with participation
* Severe pain of the hemiparetic shoulder, arm or hand either at rest or during movement.

People for whom communication problems prevent effective use of the system, will be excluded unless they have a carer who can support them effectively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Burridge, PhD, Principal Investigator — Professor at University of Southampton
Locations (1):
- University of Southampton, Southampton, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LifeCIT | Standard Care
Started | 11 | 8
Completed | 9 | 7
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LifeCIT | Standard Care | Total
Number analyzed (Participants) | 9 | 7 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.6 (19.7) | 63 (13.2) | 57.8 (16.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 5 | 6 | 11
Region of Enrollment [Number; unit: participants]
  United Kingdom | 9 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Change in Upper Limb Impairment: Motor Activity Log (MAL) Amount of Use (AOU)
Description: The MAL comprises 28 functional items, (e.g. picking up a glass; turning a key to open the door) each item is assessed by self-report on a six-point ordinal scale (0-5). Participants are asked to rate the amount of use of their hemiplegic arm for each item. Zero is scored if they have not used their affected arm, five is scored when they use their affected as often as before their stroke occurred. The final MAL score is calculated as a mean score of the individual items. The minimum and maximum mean scores are 0-5, with higher values representing better outcomes.
Time Frame: Baseline, Post intervention (three weeks) and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LifeCIT | Standard Care
Number analyzed (Participants) | 9 | 7
units on a scale
  MAL AOU baseline to three weeks | 1.02 (0.49) | 0.06 (0.42)
  MAL AOU baseline to six months | 0.60 (0.81) | 0.29 (0.45)

2. Primary Outcome: Change From Baseline in Upper Limb Impairment: Motor Activity Log (MAL) Quality of Use (QOU)
Description: he MAL comprises 28 functional items, (e.g. picking up a glass; turning a key to open the door) each item is assessed by self-report on a six-point ordinal scale (0-5). Participants are asked to rate the quality of use of their hemiplegic arm for each item. Zero is scored if they can not use their affected arm, five is scored when they can use their affected arm as well as before their stroke occurred. The final MAL score is calculated as a mean score of the individual items. The minimum and maximum mean scores are 0-5, with higher values representing better outcomes.
Time Frame: Baseline, Post Intervention (three weeks) and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LifeCIT | Usual Care
Number analyzed (Participants) | 9 | 7
units on a scale
  MAL QOU change from baseline to three weeks | 1.02 (0.5) | 0.26 (0.21)
  MAL QOU change from baseline to six months | 0.6 (0.78) | 0.23 (0.5)

3. Secondary Outcome: Change in Upper Limb Function: Wolf Motor Function Test (WMFT) Functional Ability Scale (FAS)
Description: The modified WMFT is a valid, widely used measure that scores performance of activities of daily living in a controlled and structured environment he test has 17 items which test a range of functional upper limb tasks (for example turning a key in a lock, folding a towel, retrieving a weight). Each item is scored by the time taken to complete the task, the weight lifted or hand strength as measured by a hand held goniometer. Each item is subsequently scored on a rating scale 'The Functional Ability Scale' (FAS) from 0-5. Zero is scored if the participant does not attempt the task with their hemiplegic arm, and five is scored if the task is completed with a normal movement. The mean score of all items results with a mean FAS score.
Time Frame: Baseline, Post intervention (three weeks), 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LifeCIT | Standard Care
Number analyzed (Participants) | 9 | 7
units on a scale
  WMFT FAS change from baseline to three weeks | 0.35 (0.22) | 0.02 (0.21)
  WMFT FAS change from baseline to six months | 0.30 (0.47) | 0.01 (0.36)

4. Secondary Outcome: Change in Upper Limb Impairment: Fugel Myer Upper Extremity (FMUE)
Description: The upper extremity domain of the Fugel Myer is a 0-66 point clinical assessed scale where separate Items are scored on a 3-point ordinal scale:
  0 = cannot perform, 1 = performs partially, 2 = performs fully. A higher score indicates indicates an increased level of function.
Time Frame: Baseline, Post Intervention (three weeks) and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LifeCIT | Usual Care
Number analyzed (Participants) | 9 | 7
units on a scale
  FMUE change from baseline to three weeks | 5.67 (4.42) | 2.29 (3.77)
  FMUE change from baseline to six months | 5.29 (2.43) | 4.00 (3.46)

5. Secondary Outcome: Change in Occupational Performance: Canadian Occupational Performance Measure Performance (COPM)
Description: The Canadian Occupational Performance Measure (COPM) is an individualized client-centered measure designed for use by therapists to detect a change in a client's self-perception of occupational performance over time. The COPM involves a 5-step process within a semi-structured interview conducted by a therapist. The Interview focuses on identifying activities within each performance domain that the client wants, needs, or is expected to perform. They are then asked to rate their performance and satisfaction from 0-10 for each activity identified. A score of 0 indicates they are unable to perform the activity and a score of 10 means they can complete the activity. The same scoring system is used for the COPM Satisfaction assessment with scores ranging from 0-10 and higher scores indicating greater satisfaction.
Time Frame: Baseline, Post intervention (three weeks) and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LifeCIT | Usual Care
Number analyzed (Participants) | 9 | 7
units on a scale
  COPM Performance change baseline to three weeks | 1.07 (1.19) | 0.77 (1.32)
  COPM Performance change baseline to six months | 1.69 (1.63) | 1.24 (2.35)
  COPM Satisfaction change baseline to three weeks | 1.27 (1.38) | 1.34 (1.62)
  COPM Satisfaction change baseline to six months | 1.80 (1.74) | 1.72 (1.72)

ADVERSE EVENTS:
Arm/Group | LifeCIT | Standard Care
Serious Adverse Events (participants affected / at risk) | 1/11 | 1/8
Other Adverse Events (participants affected / at risk) | 0/11 | 1/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LifeCIT (N=11) | Standard Care (N=8)
Hip fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Participant fell off side of bed before starting LifeCIT intervention - unrelated
Second stroke (Nervous system disorders) | 0 (0) | 1 (1) — Participant experienced stroke symptoms and was re-admitted to hospital
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LifeCIT (N=11) | Standard Care (N=8)
Frozen Shoulder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No